CLINICAL TRIAL: NCT06898892
Title: Comparison of the Accuracy of Fetal Weight Estimation Between Sonographic Vs. Magnetic Resonance Assessment
Brief Title: Comparison of Sonographic and MRI Weight Estimation in Fetuses with Suspected Macrosomia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Head of Maternal Fetal Medicine Unit, Western Galilee Hospital-Nahariya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0249-24-NHR; Galilee medical center (Other: Bar Ilan University)
Record Dates: First submitted 2025-02-14; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Accuracy of Sonographic Vs MRI Fetal Weight Estimation
Keywords: fetal weight estimation, accuracy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- suspected macrosomia (Experimental): suspected macrosomia at term who will undergo sonographic and MRI fetal weight estimation
  Interventions: Diagnostic Test: Fetal MRI

INTERVENTIONS:
Diagnostic Test: Fetal MRI — all participant will undergo MRI fetal weight estimation

SUMMARY:
The goal of this clinical trial is to compare the accuracy of sonographic vs. magnetic resonance fetal weight estimation in suspected fetal macrosomia in term pregnancy.

Pregnant patient at term with suspected macrosomia will participate and undergo both sonographic and magnetic resonance fetal weight estimations and the actual birthweight will be recorded and compared with the fetal weight estimations

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare the accuracy of sonographic vs. magnetic resonance fetal weight estimation in suspected fetal macrosomia in term pregnancy.

Pregnant patient at term with suspected macrosomia will participate and undergo both sonographic and magnetic resonance fetal weight estimations and the actual birthweight will be recorded and compared with the fetal weight estimations inclusion criteria: singleton pregnancies at term, suspected fetal macrosomia (>4000 gr in non GDM and >3800 gr. in GDM cases exclusion criteria-fetal anomaly, PPROM, multiple gestation The radiologist and the sonographer will be blinded to the fetal weight estimation and to the other estimation done

ELIGIBILITY:
Inclusion Criteria:

singleton pregnancy at term, suspected fetal macrosomia,

Exclusion Criteria:

* fetal anomaly multiple pregnancy PROM

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 80 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-02-13 (Estimated); Study Completion 2028-02-13 (Estimated)

PRIMARY OUTCOMES:
MRI fetal weight estimation accuracy | from enollment to Performing the MRI at 1 week
  gram

CONTACTS AND LOCATIONS:
Overall Officials: Amal shahin, Principal Investigator — Galilee Medical Center
Locations (1):
- Galilee medical center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Langer O, Berkus MD, Huff RW, Samueloff A. Shoulder dystocia: should the fetus weighing greater than or equal to 4000 grams be delivered by cesarean section? Am J Obstet Gynecol. 1991 Oct;165(4 Pt 1):831-7. doi: 10.1016/0002-9378(91)90424-p. PMID 1951539
- [Background] Kadji C, Cannie MM, Kang X, Carlin A, Benjou Etchoua S, Resta S, Dutemeyer V, Abi-Khalil F, Mazzone E, Bevilacqua E, Jani JC. Fetal magnetic resonance imaging at 36 weeks predicts neonatal macrosomia: the PREMACRO study. Am J Obstet Gynecol. 2022 Feb;226(2):238.e1-238.e12. doi: 10.1016/j.ajog.2021.08.001. Epub 2021 Aug 4. PMID 34358479
- [Background] Malin GL, Bugg GJ, Takwoingi Y, Thornton JG, Jones NW. Antenatal magnetic resonance imaging versus ultrasound for predicting neonatal macrosomia: a systematic review and meta-analysis. BJOG. 2016 Jan;123(1):77-88. doi: 10.1111/1471-0528.13517. Epub 2015 Jul 29. PMID 26224221